CLINICAL TRIAL: NCT02244814
Title: Randomized Trial of Diet in Gestational Diabetes Mellitus: Metabolic Consequences to Mother and Offspring
Brief Title: Trial of Diet in Gestational Diabetes Mellitus: Metabolic Consequences to Mother and Offspring
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-1358
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Gestational Diabetes Mellitus
Keywords: glucose; insulin resistance; dietary carbohydrate; dietary fat; adiposity; Air displacement plethysmography; Dual X-ray Absorptiometry; continuous glucose monitoring
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance; Obesity | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Choosing Healthy Options in Carbohydrate Energy (Experimental): 60% carbohydrate/25% fat/15% protein diet
  Interventions: Behavioral: Low Carbohydrate/Conventional; Behavioral: Choosing Healthy Options in Carbohydrate Energy
- Low Carbohydrate/Conventional (Active Comparator): 40% carbohydrate/45% fat/15% protein
  Interventions: Behavioral: Low Carbohydrate/Conventional; Behavioral: Choosing Healthy Options in Carbohydrate Energy

INTERVENTIONS:
Behavioral: Low Carbohydrate/Conventional — Lower-carbohydrate/conventional diet (usual care)
Behavioral: Choosing Healthy Options in Carbohydrate Energy — Choosing Healthy Options in Carbohydrate Energy

SUMMARY:
The rapidly rising risk of gestational diabetes pregnant women demands that an effective diet strategy be developed due to the high risk of fetal overgrowth, which places the newborn at increased risk for childhood obesity and metabolic syndrome. The aims of this randomized clinical trial are to compare the effects of an 8-wk isocaloric higher complex carbohydrate/lower fat diet vs. a conventional lower carbohydrate (higher fat) diet on glycemic and lipid profiles, maternal insulin resistance, placenta nutrient transporters, the maternal microbiome, neonatal intrahepatic fat, and neonatal total adiposity (primary outcome). The investigators will then follow the infants for 1-yr and measure maternal breast milk and infant microbiome composition to observe if they impact net fat mass gain differently in infants exposed to one diet vs. the other. Identifying a diet for gestational diabetes mellitus women that can effectively alter maternal/fetal metabolism is critical to reducing short- and long-term metabolic risk in this growing cohort of mothers and infants and has the potential to be applicable to overweight/obese pregnant women.

DETAILED DESCRIPTION:
The rapidly rising incidence of gestational diabetes mellitus in overweight/obese pregnant women demands that an effective diet strategy be developed due to the high risk of fetal overgrowth, which places the newborn at increased risk for childhood obesity and metabolic syndrome. However, the lack of adequate controlled randomized clinical trials for treatment of gestational diabetes with diet has resulted in consensus panels abandoning any specific diet recommendation. If effective, diet therapy has the potential to avoid the high costs of medical treatment and intensified fetal monitoring for this growing population. Although a low carbohydrate diet has historically been advocated to decrease glucose excursions after meals, carbohydrate has typically been replaced by higher fat which has been shown in animal and non-human primate data to promote insulin resistance, glucose intolerance, and liver fat deposition in the offspring. In fact, recent human data suggest that high maternal triglycerides and free fatty acids, variables sensitive to dietary manipulation, may be at least as important as glucose in contributing to excess fetal growth and infant adiposity. Preliminary data based on an R21, show that compared to a conventional lower-carbohydrate (higher in fat) diet, providing a higher complex carbohydrate (lower fat) diet effectively blunts postprandial glucose and improves fasting glucose and insulin after 6-7 weeks, with less adiposity in the newborn. The investigators global hypothesis is that compared to 8 weeks of a low-carbohydrate/higher fat diet, a higher complex carbohydrate/lower fat diet will blunt maternal post-prandial free fatty acids and improve insulin resistance. Improved insulin sensitivity will reduce fetal over-nutrition by decreasing substrate availability and down-regulating placental nutrient transporters, thereby reducing neonatal adiposity (primary outcome).This proposal builds on the investigators R21 study, which is the first randomized clinical trial to provide all meals from the time of gestational diabetes diagnosis throughout the remainder of pregnancy. The aims of this randomized trial are to compare the effects of an 8-wk isocaloric higher complex carbohydrate/lower fat diet (60% carbohydrate/25% fat) vs. a conventional low-carbohydrate (higher fat)(40% carbohydrate/45% fat) diet on maternal insulin resistance, placental nutrient transporters, and neonatal fat development. Innovative approaches by the investigators skilled multidisciplinary team include: maternal insulin resistance systemically (oral glucose tolerance Index) and locally (adipose tissue lipolysis); intestinal microbiome (transferred to the newborn); and neonatal intrahepatic fat (magnetic resonance spectroscopy). Persistence of neonatal adiposity is relevant to understanding obesity risk in these infants. As the investigators pilot data suggest infant microbiome and breast milk composition impact fat accrual after birth, the investigators will follow the infants through 1-yr of life accounting for these variables. Identifying a diet for gestational diabetes that can effectively alter maternal/fetal metabolism in late pregnancy when fetal growth accelerates is critical to reducing short- and long-term metabolic risk in this growing cohort of mothers and infants. The study results could lead to a paradigm shift for diet therapy in gestational diabetes, with potential widespread application to pregnancies affected by obesity alone.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women will be between the ages of 20-36 yrs
* BMI of 26-39 kg/m2 at the time of diagnosis
* singleton pregnancy
* no oral hypoglycemic therapy before entering the study
* diagnosed with Gestational diabetes according to the criteria established by the American College of Obstetricians and Gynecologists, specifically, they will have 2 abnormal values on a 100-g 3 hr glucose tolerance test 205, 206: Fasting>95 mg/dL but <105 mg/dL; 1hr> 180 mg/dL; 2 hr>155 mg/dL; 3 hr>140 mg/dL.

Exclusion Criteria:

* extreme hypertriglyceridemia
* overt diabetes
* suspected preexisting diabetes (A1C≥6.5%, Fasting glucose>125 mg/dL, or random glucose >200/mg/dL)
* women highly likely to fail diet by any of the following criteria will be excluded:1) Fasting glucose >105 mg/dL, due to the higher likelihood of failing diet and requiring medical treatment 139; 2) Fasting triglyceride > 400 mg/dL.
* non-English speaking
* Smokers (leading cause of low birth weight)
* Risk factors for placental insufficiency (hypertension, renal disease, thrombophilias, rheumatologic disease, preeclampsia, steroid use, history of pancreatitis, infectious disease, or intrauterine growth restriction)
* History of pancreatitis
* History of pre-term labor
* Taking beta blockers/glucocorticoids

Max Age: 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Neonatal adiposity | 5-7 days after birth
  Air-displacement plethysmography

SECONDARY OUTCOMES:
Maternal Insulin Resistance | 36 wks gestation
  Between-diet difference in post-prandial free fatty acid area-under-the-curve as a surrogate for insulin resistance
Placental fatty acid transporter protein-2 expression | Delivery
  Between diet-difference in protein expression of placental fatty acid transporter protein-2.

OTHER OUTCOMES:
Oral glucose tolerance test | Baseline, 36 wks
  75g oral glucose tolerance test; calculated Index to assess diet-induced differences in maternal insulin resistance.
Adipose Tissue Lipolysis | Baseline, 36 wks
  Diet-induced difference in adipose tissue lipolysis.
Infant Adiposity | Birth-12 mos
  Infant adiposity (air displacement plethysmography, anthropometry) from delivery - 1 year (dual x-ray absorptiometry)

CONTACTS AND LOCATIONS:
Overall Officials: Teri L Hernandez, PhD, RN, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado/Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez TL, Van Pelt RE, Anderson MA, Daniels LJ, West NA, Donahoo WT, Friedman JE, Barbour LA. A higher-complex carbohydrate diet in gestational diabetes mellitus achieves glucose targets and lowers postprandial lipids: a randomized crossover study. Diabetes Care. 2014;37(5):1254-62. doi: 10.2337/dc13-2411. Epub 2014 Mar 4. PMID 24595632